CLINICAL TRIAL: NCT06701474
Title: Association Between Phase Angle and Functional Recovery After Total Knee Arthroplasty
Brief Title: Comparison of Functional Recovery After Total Knee Arthroplasty Between Low Phase Angle and High Phase Angle Group
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 9-2024-0150
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: total knee arthroplasty; phase angle; sarcopenia; bioelectrical impedance
MeSH Terms: conditions — Osteoarthritis, Knee; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high PhA: * Patients diagnosed with knee osteoarthritis and scheduled for total knee arthroplasty.
  * Among these, patients are classified into the high PhA group if their preoperative PhA is above 4.95 for males or 4.35 for females
- low PhA: * Patients diagnosed with knee osteoarthritis and scheduled for total knee arthroplasty.
  * Among these, patients are classified into the low PhA group if their preoperative PhA is below 4.95 for males or 4.35 for females

SUMMARY:
The goal of this observational study is to compare the functional outcome of patients with end-stage knee osteoarthritis (OA) before and after total knee arthroplasty based on the phase angle level.

The main questions it aims to answer are:

* Do patients with low phase angle show worse functional recovery after total knee arthroplasty compared to those with high phase angle?
* Is postoperative physical function associated with preoperative phase angle level?

Researchers will compare postoperative physical function and muscle strength between the low and high phase angle groups to determine whether a low phase angle is associated with poorer functional recovery.

Participants will:

Perform physical function tests, isokinetic strength assessments, and bioelectrical impedance analysis before and three months after surgery.

DETAILED DESCRIPTION:
After obtaining informed consent, a pre-surgical screening is conducted. Participants complete a history survey, a sarcopenia questionnaire, and the International Physical Activity Questionnaire (IPAQ).

The screening includes a comprehensive evaluation of baseline symptoms, followed by functional assessments that incorporate bioelectrical impedance analysis, muscle strength testing, and performance-based tests:

* A modified Charlson Comorbidity Index (CCI) is used to assess comorbidity burden, and a Numeric Pain Rating Scale (NPRS) records participants' initial pain levels.
* Radiographic assessments are performed to evaluate the frontal alignment of the lower extremities and the radiographic severity of knee osteoarthritis (OA) using the Kellgren-Lawrence (K-L) grading system.
* Multifrequency bioelectrical impedance analysis (BIA) is used to measure phase angle and body composition.
* Handgrip strength is measured through three trials on each side, with the average recorded.
* Knee strength is measured using an isokinetic dynamometer.
* Performance-based tests include the 10-meter walk test, the Timed Up and Go (TUG) test, and the Berg Balance Scale (BBS).

Follow-up assessments are conducted three months after total knee arthroplasty, with participants undergoing the same protocol for performance-based tests, isokinetic knee strength evaluation, and bioelectrical impedance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 55 and over (based on the age on their national ID at the time of consent)
* Individuals diagnosed with knee OA based on medical history, physical examination, and radiographic assessments.
* Individuals who plan to perform total knee arthroplasty

Exclusion Criteria:

* Individuals with gait disturbance due to neurologic disorders such as Parkinson disease, stroke and dementia
* Individuals with severe cardiac, pulmonary, or musculoskeletal disorders that limited quadriceps strength and physical function
* Individuals with knee osteoarthritis due to secondary causes such as rheumatic or traumatic arthritis
* Individuals with a history of any knee surgery within one year.
* Individuals considered clinically unsuitable for the study by the researchers or person in charge based on significant medical findings.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single general hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-09-23 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | Baseline and 3 months after surgery
  Researchers ask patients to rise from a seated position, walk a distance of 3 m, turn around, return to the chair, and sit back.
  The average time of three trials was recorded as a result
10 meter walk test (10MWT) | Baseline and 3 months after surgery
  Patients are instructed to walk 14 m, including 2 m at both ends for acceleration and deceleration, at their comfortable speed.
  Gait speed was calculated by dividing the 10m distance by the time taken.
Berg balance scale (BBS) | Baseline and 3 months after surgery
  Patients are asked to perform 14 tasks regarding the static and dynamic balance of patients. Each task was rated on a five-point scale from 0 to 4, with a total score of 56.

SECONDARY OUTCOMES:
Isokinetic peak torque of knee flexion at 60°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the peak flexion torque is performed at preset constant angular velocities, 60°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic peak torque of knee flexion at 150°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the peak flexion torque is performed at preset constant angular velocities, 150°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic peak torque of knee extension at 60°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the peak extension torque is performed at preset constant angular velocities, 60°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic peak torque of knee extension at 150°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the peak extension torque is performed at preset constant angular velocities, 150°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic total work of knee flexion at 60°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the total knee flexion effort is performed at preset constant angular velocities, 60°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic total work of knee flexion at 150°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the total knee flexion effort is performed at preset constant angular velocities, 150°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic total work of knee extension at 60°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the total knee extension effort is performed at preset constant angular velocities, 60°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Isokinetic total work of knee extension at 150°/s | Baseline and 3 months after surgery
  * Isokinetic knee assessment is assessed using an isokinetic dynamometer (Cybex NORM®, Humac, CA, USA).
  * Each participant is positioned on an adjustable chair and secured to the equipment with straps across the trunk, hip, and thigh.
  * Gravity correction measurements are made according to the manufacturer's instructions.
  * Participants are instructed on standardized procedures before and during the test.
  * Concentric measurement of the total knee extension effort is performed at preset constant angular velocities, 150°/s, with a rest period between each trial to prevent fatigue and ensure consistent effort levels.
  * Participants warm up with five to six submaximal practice repetitions before each test series. After repeating three times, the examiner records the average value.
Whole body phase angle at 50kHz | Baseline and 3 months after surgery
  * Whole body phase angle is calculated using the multifrequency Bioelectrical impedance analysis (BIA) with the InBody S10 (BioSpace, Seoul, Korea).
  * Before measurement, all patients are asked to fast for a minimum of 3 hours with the bladder emptied and avoid alcohol or vigorous activity.
  * Tetrapolar 8-point electrodes are placed on the dorsal surfaces of both wrist and foot according to the manufacturer's instruction.
  * After resting for 15 minutes, a weak current under 100uA is applied to measure the reactance (Xc) and impedance (R) of 6 Different Frequencies (1kHz, 5kHz, 50kHz, 250kHz, 500kHz, 1000kHz).
  * A whole body Phase angle is calculated as an arctangent of the Xc to R ratio at 50kHz. [Phase angle (degrees) arctan(Xc/R) (180/π)]

CONTACTS AND LOCATIONS:
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uemura K, Doi T, Tsutsumimoto K, Nakakubo S, Kim MJ, Kurita S, Ishii H, Shimada H. Predictivity of bioimpedance phase angle for incident disability in older adults. J Cachexia Sarcopenia Muscle. 2020 Feb;11(1):46-54. doi: 10.1002/jcsm.12492. Epub 2019 Aug 22. PMID 31436391
- [Result] Martins PC, Alves Junior CAS, Silva AM, Silva DAS. Phase angle and body composition: A scoping review. Clin Nutr ESPEN. 2023 Aug;56:237-250. doi: 10.1016/j.clnesp.2023.05.015. Epub 2023 Jun 1. PMID 37344079
- [Result] Stapel SN, Looijaard WGPM, Dekker IM, Girbes ARJ, Weijs PJM, Oudemans-van Straaten HM. Bioelectrical impedance analysis-derived phase angle at admission as a predictor of 90-day mortality in intensive care patients. Eur J Clin Nutr. 2018 Jul;72(7):1019-1025. doi: 10.1038/s41430-018-0167-1. Epub 2018 May 11. PMID 29748659
- [Result] Sardinha LB, Rosa GB. Phase angle, muscle tissue, and resistance training. Rev Endocr Metab Disord. 2023 Jun;24(3):393-414. doi: 10.1007/s11154-023-09791-8. Epub 2023 Feb 10. PMID 36759377
- [Result] Harris IA, Harris AM, Naylor JM, Adie S, Mittal R, Dao AT. Discordance between patient and surgeon satisfaction after total joint arthroplasty. J Arthroplasty. 2013 May;28(5):722-7. doi: 10.1016/j.arth.2012.07.044. Epub 2013 Feb 23. PMID 23462496
- [Result] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Result] Capin JJ, Bade MJ, Jennings JM, Snyder-Mackler L, Stevens-Lapsley JE. Total Knee Arthroplasty Assessments Should Include Strength and Performance-Based Functional Tests to Complement Range-of-Motion and Patient-Reported Outcome Measures. Phys Ther. 2022 Jun 3;102(6):pzac033. doi: 10.1093/ptj/pzac033. PMID 35358318
- [Result] Wieczorek M, Rotonda C, Guillemin F, Rat AC. What Have We Learned About the Course of Clinical Outcomes After Total Knee or Hip Arthroplasty? Arthritis Care Res (Hoboken). 2020 Nov;72(11):1519-1529. doi: 10.1002/acr.24045. PMID 31421025
- [Result] GBD 2021 Osteoarthritis Collaborators. Global, regional, and national burden of osteoarthritis, 1990-2020 and projections to 2050: a systematic analysis for the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 Aug 21;5(9):e508-e522. doi: 10.1016/S2665-9913(23)00163-7. eCollection 2023 Sep. PMID 37675071